CLINICAL TRIAL: NCT01654224
Title: Randomized Trial of High Dose Influenza Vaccine in Long Term Care Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, David Nace, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO10110247
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Influenza
Keywords: Influenza in Long Term Care Setting; High dose Inactivated influenza vaccine; Standard dose inactivated influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Inactivated Influenza Vaccine (Active Comparator): For HDIV,0.5 ml of high dose inactivated influenza vaccine consisting of a total of 180mcg (60 mcg each strain) of influenza virus hemagglutinin
  Interventions: Biological: High Dose Inactivated Influenza Vaccine
- Standard Dose Inactivated Influenza Vaccine (Active Comparator): For SDIV, 0.5 ml of standard dose inactivated influenza vaccine consisting of a total of 45 mcg (15 mcg of each strain) of influenza virus hemagglutinin
  Interventions: Biological: Standard Dose Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: High Dose Inactivated Influenza Vaccine — 0.5 ml HDIV consisting of 180 mcg (60 mcg each strain) of influenza virus hemagglutinin
  Arms: High Dose Inactivated Influenza Vaccine
Biological: Standard Dose Inactivated Influenza Vaccine — 0.5 ml of standard dose inactivated influenza vaccine consisting of a total of 45 mcg (15 mcg each strain) of influenza virus hemagglutinin
  Arms: Standard Dose Inactivated Influenza Vaccine

SUMMARY:
The purpose of the study is to compare the performance of two currently available influenza (flu) vaccines. This study will try and determine if the high dose flu vaccine provides protection that is the same or better than that of regular dose flu vaccine. Both the regular dose and the high dose flu vaccines are approved by the FDA for use in older adults.

DETAILED DESCRIPTION:
Influenza and pneumonia are the fifth leading cause of death in the United States, the leading cause of vaccine preventable death, and the leading cause of infection related deaths among nursing home residents(Nace, Drinka et al.2010). Each year, an estimated 36,000 individuals die from seasonal influenza and over 90% of these deaths occur among older adults, primarily the frail older adults residing in LTC settings(Fiore,Uyeki et al. 2010).Vaccination is the most effective means of preventing influenza (Nichol and Treanor 2006). Despite increasing success in immunizing LTC residents though, outbreaks continue to occur annually with case fatality rates ranging between 5-55% (Nace 2008). Older adults have a reduced response to influenza vaccination, in part due to age related immunosenescence (Keitel, Atmar et al. 1121; Skowronski, Tweed et al. 2008). It is widely recognized that more effective vaccine options are needed for frail older adults. One option is to increase the hemagglutinin (HA) dose in influenza vaccines in an effort to increase antibodies to hemagglutinin. To date, no studies have evaluated the effectiveness of the HDIV among LTC residents.

ELIGIBILITY:
Inclusion Criteria:

* Residents of one of the participating LTC sites
* 65 years or older at the time of consent
* require assistance in two or more Instrumental Activities of Daily Living and/or one or more Activities of Daily Living as identified by facility staff

Exclusion Criteria:

* Age less than 65 years
* Life expectancy less than 6 months
* History of allergic reaction to influenza vaccine, its components, or eggs
* History of severe allergic reaction to latex
* History of Guillian-Barre Syndrome
* Actively undergoing chemotherapy
* Actively undergoing radiation therapy
* Use of prednisone (or other steroid) at prednisone-equivalent dosages of 10mg or higher within the past 14 days
* Serious current immunosuppression or immunosuppression expected in the next 6 weeks
* Any condition that, in the opinion of the investigator,might interfere with the evaluation of study objectives

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Nace, MD, MPH, CMD, Principal Investigator — University of Pittsburgh, Division of Geriatric Medicine
Locations (1):
- University of Pittsburgh, Division of Geriatric Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Nace DA, Lin CJ, Ross TM, Saracco S, Churilla RM, Zimmerman RK. Randomized, controlled trial of high-dose influenza vaccine among frail residents of long-term care facilities. J Infect Dis. 2015 Jun 15;211(12):1915-24. doi: 10.1093/infdis/jiu622. Epub 2014 Dec 17. PMID 25525051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled during the 2011-2012 and 2012-2013 influenza seasons
Pre-assignment Details: A total of 205 participants from 15 community-based LTCFs who met all inclusion and none of the exclusion criteria were enrolled.
Groups:
- HD IIV: Frail adults 65 years or older who received Fluzone High Dose intramuscularly.
- SD IIV: Frail adults 65 years or older who received Fluzone Standard Dose intramuscularly
Period: Overall Study
Arm/Group | HD IIV | SD IIV
Started | 95 | 110
Completed | 89 | 98
Not Completed | 6 | 12
Not completed — Lost to Follow-up | 2 | 2
Not completed — Did not receive allocation | 1 | 8
Not completed — Insufficient blood sample | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- HD IIV: Frail adults 65 years and older who received Fluzone High Dose intramuscularly
- SD IIV: Frail adults 65 years and older who received Fluzone Standard Dose intramuscularly
- Total: Total of all reporting groups
Arm/Group | HD IIV | SD IIV | Total
Number analyzed (Participants) | 89 | 98 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 89 | 98 | 187
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 71 | 128
  Male | 32 | 27 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 89 | 96 | 185
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 89 | 96 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 89 | 98 | 187

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of High-dose Inactivated Influenza Vaccine(HDIV) Versus Standard Dose Inactivated Influenza Vaccine(SDIV) Among Residents of Long Term Care(LTC) Settings
Description: The primary objective of this study is to determine the noninferiority of high- dose inactivated influenza vaccine (HDIV) versus standard dose inactivated influenza vaccine(SDIV)among residents of long term care(LTC)settings.Non-inferiority will be determined by comparing baseline and one month post vaccination HAI and MN titers using non-inferiority analysis.
Time Frame: 30 days
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | High Dose Inactivated Influenza Vaccine | Standard Dose Inactivated Influenza Vaccine
Number analyzed (Participants) | 89 | 98
titers
  A/California/07/2009(H1N1)-2011-2012 Season | 78.2 [45.1 to 135.7] | 27.4 [17 to 44.3]
  A/Victoria/210/2009(H3N2 | 26.2 [17.1 to 40.0] | 10.2 [7.0 to 14.8]
  B/Brisbane/60/2008 | 25.6 [18.7 to 34.9] | 14.3 [11.1 to 18.4]
  A/California/07/2009(H1N1)- 2012-2013 Season | 45.6 [32.9 to 63.2] | 50.0 [37.4 to 67]
  A/Victoria/361/2011(H3N2) | 23.4 [17.6 to 31] | 14.2 [11.0 to 18.4]
  B/Texas/6/2011 | 26.0 [21.2 to 31.9] | 17.4 [13.9 to 21.9]
Statistical Analysis 1: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — An upper bound >0.67 of the 2-sided 95% CI of the ratio of postvaccination GMTHD to GMTSD indicated noninferiority. A lower bound of ≥1.0 of the 2-sided 95% CI of the ratio of GMTHD to GMTSD indicated superiority; p = .005, t-test, 2 sided — A/California/07/2009(H1N1)
Statistical Analysis 2: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .001, t-test, 2 sided — A/Victoria/210/2009(H3N2)
Statistical Analysis 3: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .004, t-test, 2 sided — B/Brisbane/60/2008
Statistical Analysis 4: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .672, t-test, 2 sided — A/California/07/2009(H1N1)
Statistical Analysis 5: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .011, t-test, 2 sided — A/Victoria/361/2011(H3N2)
Statistical Analysis 6: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .010, t-test, 2 sided — B/Texas/6/2011

2. Secondary Outcome: Non-inferiority and Immunoprotection Persistence at 6 Months
Description: Compare the immunogenicity via HAI and MN titers for HDIV and SDIV at 6 months in frail LTC residents
Time Frame: 6 months
Population: The above numbers reflect the participants with data available at 6 months. Eleven subjects (five in the high dose and 6 in the standard dose groups) died of non-related causes. Some of the samples were insufficient or unable to be collected.
Measure: Geometric Mean (90% Confidence Interval); unit: Titers
Arm/Group | High Dose Inactivated Influenza Vaccine | Standard Dose Inactivated Influenza Vaccine
Number analyzed (Participants) | 79 | 83
Titers
  A/California/07/2009(H1N1) 2011-2012 Season | 59.7 [33.5 to 106.3] | 28.3 [15.3 to 52.4]
  A/Victoria/210/2009(H3N2) | 22.3 [14.5 to 34.3] | 9.4 [6 to 14.8]
  B/Brisbane/60/2008 | 22.9 [16.3 to 32] | 15.4 [11.8 to 20.2]
  A/California/07/2009(H1N1) @012-2013 Season | 46.8 [33.2 to 65.9] | 51.8 [37.8 to 71.1]
  A/Victoria/361/2011(H3N2) | 24.7 [18.3 to 33.2] | 13.4 [10.3 to 17.5]
  B/Texas/6/2011 | 25.3 [20.8 to 30.9] | 18.9 [14.9 to 23.9]
Statistical Analysis 1: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .074, t-test, 2 sided — A/California/07/2009(H1N1)
Statistical Analysis 2: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .006, t-test, 2 sided — A/Victoria/210/2009(H3N2)
Statistical Analysis 3: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .069, t-test, 2 sided — B/Brisbane/60/2008
Statistical Analysis 4: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .663, t-test, 2 sided — A/California/07/2009(H3N2)
Statistical Analysis 5: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .003, t-test, 2 sided — A/Victoria/361/2011(H3N2)
Statistical Analysis 6: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .063, t-test, 2 sided — B/Texas/6/2011

3. Primary Outcome: Non-inferiority of High-dose Inactivated Influenza Vaccine(HDIV) Versus Standard Dose Inactivated Influenza Vaccine(SDIV) Among Residents of Long Term Care(LTC) Settings
Description: as for outcome 1
Time Frame: Day 0
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | High Dose Inactivated Influenza Vaccine | Standard Dose Inactivated Influenza Vaccine
Number analyzed (Participants) | 89 | 98
titers
  A/California/07/2009(H1N1)2011-2012 Season | 17.1 [11.3 to 25.9] | 16.6 [10.3 to 26.7]
  A/Victoria/210/2009(H3N2 | 8.9 [6.5 to 12.3] | 7.3 [5.3 to 10.0]
  B/Brisbane/60/2008 | 15.3 [10.3 to 22.6] | 11.6 [8.6 to 15.5]
  A/California/07/2009(H1N1) 2012-2013 Season | 23.6 [16.7 to 33.4] | 32.3 [23.8 to 43.9]
  A/Victoria/361/2011(H3N2) | 7.2 [6.1 to 8.3] | 6.2 [5.4 to 7.1]
  B/Texas/6/2011 | 7.9 [6.5 to 9.5] | 9.1 [7.5 to 11]
Statistical Analysis 1: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .917, t-test, 2 sided — A/California/07/2009(H1N1)
Statistical Analysis 2: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .360, t-test, 2 sided — A/Victoria/210/2009(H3N2)
Statistical Analysis 3: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .248, t-test, 2 sided — B/Brisbane/60/2008
Statistical Analysis 4: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .178, t-test, 2 sided — A/California/07/2009(H1N1)
Statistical Analysis 5: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .152, t-test, 2 sided — A/Victoria/361/2011(H1N2)
Statistical Analysis 6: Comparison: High Dose Inactivated Influenza Vaccine vs Standard Dose Inactivated Influenza Vaccine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .285, t-test, 2 sided — B/Texas/6/2011

ADVERSE EVENTS:
Arm/Group | HD IIV | SD IIV
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/98
Other Adverse Events (participants affected / at risk) | 0/89 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No